CLINICAL TRIAL: NCT05012657
Title: Validation of Point Partial User Needs With Partial Finger Amputees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Point Designs (Industry)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 299089
Record Dates: First submitted 2021-08-12; First posted 2021-08-19 (Actual); Results first posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-08

CONDITIONS: Amputation; Traumatic, Hand

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Prosthesis (Experimental): Patient is temporarily fit with Point Partial partial finger prosthetic system
  Interventions: Device: Point Partial

INTERVENTIONS:
Device: Point Partial — The Point Partial partial finger prosthetic system consists of 1-4 ratcheting mechanical partial digits and mounting brackets

SUMMARY:
The objective of the device feasibility study will be to validate the user needs of the Point Partial system. This study will be a single group intervention model where one group of 5 partial finger amputees will be asked to perform several tasks. Successful completion of a task results in a fulfilled user need. Failure to complete a task results in an unfulfilled user need.

ELIGIBILITY:
Inclusion Criteria:

* Partial finger amputees with partial absence of index and/or middle fingers and presence of thumb. Additional finger loss is acceptable if all other criterion are met.
* Fluent in English
* Individuals aged 18 or greater
* Patients may present with either fused or mobile MCP joints.

Exclusion Criteria:

* Significant cognitive deficits as determined upon clinical evaluation
* Significant neurological deficits as determined upon clinical evaluation
* Significant physical deficits of the residual limb impacting full participation in the study as determined upon clinical evaluation
* Uncontrolled pain or phantom pain impacting full participation in the study as determined upon OT evaluation
* Serious uncontrolled medical problems as judged by the project therapist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Colorado Denver | Anschutz Medical Campus, Aurora, Colorado
  - Point Designs, Lafayette, Colorado

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prosthesis
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Prosthesis
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: VAL-1: System Comfort Validation Test
Description: User wears Point Partial(s) for a full day (Pass/Fail). This validation method was used to confirm the following user need of the Point Partial has been met: Point Partial shall be comfortable for a full day's use. A simple pass/fail result was recorded for each user need for each participant. An overall passing rate above 80% across all user needs and participants is considered a success. Each participant attended a single-day experimental session. A day-use prosthetic socket was fabricated and Point Partials were mounted to the socket. Then, each participant attempted the validation test.
Time Frame: Day 1 (8 hours)
Measure: Number; unit: % of participants who Passed test
Arm/Group | Prosthesis
Number analyzed (Participants) | 5
% of participants who Passed test | 100

2. Primary Outcome: VAL-2: Unilateral Function Validation Test
Description: User flexes and extends the Point Partial(s) without using contralateral hand (Pass/Fail). This validation method was used to confirm the following user need of the Point Partial has been met: Point Partial shall allow the user to flex and extend finger without their second hand. A simple pass/fail result was recorded for each user need for each participant. An overall passing rate above 80% across all user needs and participants is considered a success. Each participant attended a single-day experimental session. A day-use prosthetic socket was fabricated and Point Partials were mounted to the socket. Then, each participant attempted the validation test.
Time Frame: Day 1 (10 minutes)
Measure: Number; unit: % of participants who Passed test
Arm/Group | Prosthesis
Number analyzed (Participants) | 5
% of participants who Passed test | 100

3. Primary Outcome: VAL-3.1: System Robustness Validation Test With 25 lb Bag
Description: User lifts a 25 lb. bag with Point Partial(s) (Pass/Fail). This validation method was used to confirm the following user need of the Point Partial has been met: Point Partial shall be robust enough to operate in challenging environments. A simple pass/fail result was recorded for each user need for each participant. An overall passing rate above 80% across all user needs and participants is considered a success. Each participant attended a single-day experimental session. A day-use prosthetic socket was fabricated and Point Partials were mounted to the socket. Then, each participant attempted the validation test.
Time Frame: Day 1 (10 minutes)
Measure: Number; unit: % of participants who Passed test
Arm/Group | Prosthesis
Number analyzed (Participants) | 5
% of participants who Passed test | 100

4. Primary Outcome: VAL-3.2: Robustness Validation Test With Hammer
Description: User grips a hammer with Point Partial(s) and drives a nail into a piece of wood (Pass/Fail). This validation method was used to confirm the following user need of the Point Partial has been met: Point Partial shall be robust enough to operate in challenging environments. A simple pass/fail result was recorded for each user need for each participant. An overall passing rate above 80% across all user needs and participants is considered a success. Each participant attended a single-day experimental session. A day-use prosthetic socket was fabricated and Point Partials were mounted to the socket. Then, each participant attempted the validation test.
Time Frame: Day 1 (10 minutes)
Measure: Number; unit: % of participants who Passed test
Arm/Group | Prosthesis
Number analyzed (Participants) | 5
% of participants who Passed test | 100

5. Primary Outcome: VAL-4: Object Release Validation Test
Description: User releases Point Partial(s) while performing an active grasp by pressing the dorsal button (Pass/Fail). This validation method was used to confirm the following user need of the Point Partial has been met: Point Partial shall be releasable while performing active grasps. A simple pass/fail result was recorded for each user need for each participant. An overall passing rate above 80% across all user needs and participants is considered a success. Each participant attended a single-day experimental session. A day-use prosthetic socket was fabricated and Point Partials were mounted to the socket. Then, each participant attempted the validation test.
Time Frame: Day 1 (10 minutes)
Measure: Number; unit: % of participants who Passed test
Arm/Group | Prosthesis
Number analyzed (Participants) | 5
% of participants who Passed test | 100

6. Primary Outcome: VAL-5: Position Function Validation Test
Description: User positions Point Partial(s) into each of the locking positions (Pass/Fail). This validation method was used to confirm the following user need of the Point Partial has been met: Point Partial shall have a smooth ratcheting mechanism. A simple pass/fail result was recorded for each user need for each participant. An overall passing rate above 80% across all user needs and participants is considered a success. Each participant attended a single-day experimental session. A day-use prosthetic socket was fabricated and Point Partials were mounted to the socket. Then, each participant attempted the validation test.
Time Frame: Day 1 (10 minutes)
Measure: Number; unit: % of participants who Passed test
Arm/Group | Prosthesis
Number analyzed (Participants) | 5
% of participants who Passed test | 100

7. Primary Outcome: VAL-6: Extension Function Validation Test
Description: User activates spring-back mechanism by using (1) contralateral hand, (2) tabletop, and (3) side or thigh throughout day without failed extension (Pass/Fail). This validation method was used to confirm the following user need of the Point Partial has been met: Point Partial shall have a reliable auto spring-back mechanism. A simple pass/fail result was recorded for each user need for each participant. An overall passing rate above 80% across all user needs and participants is considered a success. Each participant attended a single-day experimental session. A day-use prosthetic socket was fabricated and Point Partials were mounted to the socket. Then, each participant attempted the validation test.
Time Frame: Day 1 (10 minutes)
Measure: Number; unit: % of participants who Passed test
Arm/Group | Prosthesis
Number analyzed (Participants) | 5
% of participants who Passed test | 100

8. Primary Outcome: VAL-7: Grip Functions Validation Test
Description: User grips a 5 lb. cylindrical smooth object using Point Partial(s) for 10 seconds (Pass/Fail). This validation method was used to confirm the following user need of the Point Partial has been met: Point Partial shall have high grip surface friction. A simple pass/fail result was recorded for each user need for each participant. An overall passing rate above 80% across all user needs and participants is considered a success. Each participant attended a single-day experimental session. A day-use prosthetic socket was fabricated and Point Partials were mounted to the socket. Then, each participant attempted the validation test.
Time Frame: Day 1 (10 minutes)
Measure: Number; unit: % of participants who Passed test
Arm/Group | Prosthesis
Number analyzed (Participants) | 5
% of participants who Passed test | 100

9. Primary Outcome: VAL-8: Fine Motor Function Validation Test
Description: User picks up 1 coin from a smooth tabletop (Pass/Fail). This validation method was used to confirm the following user need of the Point Partial has been met: Point Partial shall have a pronounced fingernail. A simple pass/fail result was recorded for each user need for each participant. An overall passing rate above 80% across all user needs and participants is considered a success. Each participant attended a single-day experimental session. A day-use prosthetic socket was fabricated and Point Partials were mounted to the socket. Then, each participant attempted the validation test.
Time Frame: Day 1 (10 minutes)
Measure: Number; unit: % of participants who Passed test
Arm/Group | Prosthesis
Number analyzed (Participants) | 5
% of participants who Passed test | 100

10. Primary Outcome: VAL-9: Overall Function & Robustness Validation Test
Description: User performs VAL-1 through VAL-8 (Pass/Fail). This validation method was used to confirm the following user need of the Point Partial has been met: Point Partial shall be robustly attached to mounting system. A simple pass/fail result was recorded for each user need for each participant. An overall passing rate above 80% across all user needs and participants is considered a success. Each participant attended a single-day experimental session. A day-use prosthetic socket was fabricated and Point Partials were mounted to the socket. Then, each participant attempted the validation test.
Time Frame: Day 1 (8 hours)
Measure: Number; unit: % of participants who Passed test
Arm/Group | Prosthesis
Number analyzed (Participants) | 5
% of participants who Passed test | 100

ADVERSE EVENTS:
Time Frame: an average of 1 day
Arm/Group | Prosthesis
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT05012657/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-22): https://cdn.clinicaltrials.gov/large-docs/57/NCT05012657/SAP_001.pdf